CLINICAL TRIAL: NCT02636101
Title: Xamiol® Gel in BODY Psoriasis : lonG-term Management of Psoriasis vUlgARis With Xamiol® Gel in Daily Clinical Practice of Russian Dermatologists. A Long-term Observational, Prospective Study
Brief Title: Xamiol®Gel in BODY Psoriasis: A One-year Non-interventional Study
Acronym: BODYGUARD
Status: Completed | Type: Observational
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-DAIVOBETGEL-1210
Record Dates: First submitted 2015-12-09; First posted 2015-12-21 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2017-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — calcipotriene; betamethasone dipropionate, calcipotriol drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Calcipotriol/betamethasone dipropionate gel — Topical treatment of psoriasis plaques located on the body
  Other Names: Xamiol®; Daivobet®

SUMMARY:
This study aims to describe the patient population treated and the real-life patients' experiences with Xamiol®gel in the long term, up to 52 weeks management of body psoriasis vulgaris in Russia. The result will increase the knowledge on Xamiol®gel enabling dermatologists and patients to optimize its use in the long term management of psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Psoriasis vulgaris on body
* Patients planned to receive topical treatment on the body with calcipotriol/betamethasone gel
* Written informed consent

Exclusion Criteria:

* No or very mild symptoms of psoriasis vulgaris on the body at study start
* Any on-going treatments at study start with topical steroids, salicylic acid or its combination
* Other topical treatment for body psoriasis
* Pregnancy or planned pregnancy within treatment period
* Contraindications according to prescribing information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with body psoriasis who (at their physician's discretion) are eligible to receive topical treatment with calcipotriol/betamethasone gel
Sampling Method: Non-Probability Sample
Enrollment: 603 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-02-15 (Actual)

PRIMARY OUTCOMES:
Patient reported treatment satisfaction | Around 8 weeks after treatment initiation
  Patient preference compared with previous therapy
Adherence to treatment | Around 8 weeks after treatment initiation
  Number of days during the last 7 days with no treatment

SECONDARY OUTCOMES:
Physician Global Assessment of Psoriasis | Around 8 weeks after treatment initiation
Frequency of treatment after completion of initial treatment | 12 months
To evaluate the effect of treatment with Xamiol®gel on patients quality of life | Around 8 weeks
  Dermatology Life Quality Index (DLQI)
Overall rate of treatment success | Around 8 weeks
  Clear or almost clear by Physician Psoriasis Global Assessment
Patient's willingness to pay | 12 months
  Total consumption during study period in Russia where Xamiol®gel is not reimbursed

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Petrunin, MD, PhD, Study Director — LEO Pharmaceutical Products LLC
Locations (1):
- Municipal out-patient clinic 7, Saratov, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Results of the long-term observational noninterventional prospective study BODYGUARD in psoriasis patients Bakulev, A. L. [2] , and Petrunin, D. D. [1] , Vestnik dermatologii i venerologii (volume 95, issue 4, pages 87-93) , 10/19/2019
- [Result] EADV 2019 Abstract P1788. Bakulev AL, Petrunin DD. Results from a long-term, observational, non-interventional, prospective study in patients with body psoriasis based on patient-reported outcomes and physician's assessments (BODYGUARD).
- See also: Results — https://doi.org/10.25208/0042-4609-2019-95-4-87-93